CLINICAL TRIAL: NCT06604390
Title: The EFFECTS of GAMBIR CATECHIN (UNCARIA GAMBIR ROXB) SUPPLEMENTATION on COGNITIVE FUNCTION, EXPRESSION of AMYLOID PRECURSOR PROTEIN (APP), MICROTUBULE ASSOCIATED PROTEIN TAU (MAPT), BRAIN-DERIVED NEUROTROPHIC FACTOR (BDNF), INTERLEUKIN 10 (IL-10), TRANSFORMING GROWTH FACTOR-BETA (TGF-BETA), and PLASMA MALONDIALDEHYDE (MDA) LEVELS in the ELDERLY
Brief Title: The EFFECTS of GAMBIR CATECHIN (UNCARIA GAMBIR ROXB) SUPPLEMENTATION on COGNITIVE FUNCTION, EXPRESSION of APP, MAPT, BDNF, IL-10, TGF-Β GENES, and PLASMA MDA LEVELS in the ELDERLY.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rahmi Novita Yusuf (Other)
Collaborators: Andalas University (Other)
Responsible Party: Sponsor-Investigator, Rahmi Novita Yusuf, Principal Investigator, Andalas University
Organization: Andalas University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 115/UN.16.2/KEP-FK/2024; TheResearchEthicsCommittee Fac (Other: Andalas Univercity)
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Elderly Individuals Aged 60 Years or Older; Mild Cognitive Impairment (MCI)
Keywords: Catechin; Cognitive function; cognitive funtion
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Objective:
  This clinical trial aims to investigate the effects of gambir catechin supplementation on cognitive function, and plasma levels of APP, MAPT, BDNF, IL-10, TGF-beta, and MDA in the elderly.
  Research Design: A randomized controlled trial (RCT) design will be used. Population and Sample:The target population for this study is the elderly aged 60 years and above with mild cognitive impairment (MoCA-INA score of 20-25) residing in Padang City, West Sumatra, Indonesia.
  Intervention
  1. Participants will be randomly assigned to either the intervention or control group.
  2. The intervention group will receive gambier catechin supplementation (Uncaria gambir Roxb) at a daily dose of [224 mg] for 12 weeks.
  3. The control group will receive a placebo.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Catechin Group Arm 2: Placebo Group (Placebo Comparator): Arm 1: Catechin Group. Participants in this group received one capsule of gambir catechin daily, with a dosage of 224 mg.
  Arm 2: Placebo Group. Participants in this group received one placebo capsule daily, with a dosage of 224 mg.
  Interventions: Dietary Supplement: catechin extracts (health food); Other: plasebo
- Effects of Gambier Catechin Supplementation on Cognitive Function, APP, MAPT, (Experimental): Gambir purified with a minimum of 90% (+)-Catechin content. Dosage of 224 mg catechin per capsule, once daily.
  Interventions: Dietary Supplement: catechin extracts (health food); Other: plasebo

INTERVENTIONS:
Dietary Supplement: catechin extracts (health food) — Type of intervention:
  1. Purified gambir ≥ 90% (+)-Catechin
  2. Dosage of 224 mg catechin capsule, once daily
  3. Dosage of 224 mg placebo capsule, once daily
  4. Cognitive function was assessed using MoCA-Ina and gene markers APP, MAPT, BDNF, IL-10, TGF-Beta and MDA Plasma."
Other: plasebo — Dosage of 224 mg placebo per capsule, once daily. Cognitive function was assessed using the MoCA-Ina and biomarkers including APP, MAPT, BDNF, IL-10, TGF-Beta, and plasma MDA.

SUMMARY:
Objective The primary objective of this clinical trial is to investigate the effects of gambir catechin administration on cognitive function, the expression of amyloid precursor protein (APP), microtubule-associated protein tau (MAPT), brain-derived neurotrophic factor (BDNF), interleukin-10 (IL-10), transforming growth factor beta (TGF-beta), and plasma malondialdehyde (MDA) levels in elderly individuals.

Research Questions

The primary research questions to be addressed in this study are as follows:

1. Does the administration of gambir catechin (Uncaria gambir Roxb) improve cognitive function as measured by the Montreal Cognitive Assessment-Indonesia (MoCA-INA) in the elderly after 12 weeks of intervention?
2. Does the administration of gambir catechin (Uncaria gambir Roxb) affect the expression of APP, MAPT, BDNF, IL-10, and TGF-beta genes in the elderly after 12 weeks of intervention?
3. Does the administration of gambir catechin (Uncaria gambir Roxb) influence plasma MDA levels in the elderly after 12 weeks of intervention? Methodology

To answer these questions, researchers will compare the effects of gambir catechin with a placebo (an inert substance). This double-blind, randomized controlled trial will involve:

* Participant Recruitment: Elderly individuals will be recruited and randomly assigned to either the gambir catechin or placebo group.
* Intervention: Participants will receive daily doses of gambir catechin or a placebo for 12 weeks.
* Assessments: Cognitive function, gene expression, and plasma MDA levels will be assessed at baseline and after 12 weeks of intervention.
* Data Analysis: The collected data will be analyzed using appropriate statistical methods to determine the effects of gambir catechin.

Participant Involvement

Participants will be required to:

* Consume the assigned supplement (gambir catechin or placebo) daily.
* Attend regular follow-up visits at the research center.
* Report any adverse events or changes in their health during the study period.

DETAILED DESCRIPTION:
Effects of Gambier Catechin (Uncaria gambir Roxb) Supplementation on Cognitive Function, APP, MAPT, BDNF, IL-10, TGF-β Gene Expression, and Plasma MDA Levels in the Elderly

1. Background Problem: The increasing prevalence of mild cognitive impairment among the elderly and its impact on their quality of life.

   Research Gap: A lack of research on the utilization of local plants, specifically catechin, an active compound found in gambier leaves, which possesses antioxidant and anti-inflammatory properties and may enhance cognitive function in the elderly population in Indonesia.

   Research Objective: To investigate the effects of gambier catechin (Uncaria gambir Roxb) supplementation on cognitive function, APP, MAPT, BDNF, IL-10, TGF-β gene expression, and plasma MDA levels in the elderly.
2. Hypothesis

   1. There is an effect of gambier catechin (Uncaria gambir Roxb) supplementation on improving cognitive function as measured by the MoCA-INA test in the elderly after 12 weeks of supplementation.
   2. There is an effect of gambier catechin (Uncaria gambir Roxb) supplementation on decreasing the expression of APP, MAPT, TGF-β genes and increasing the expression of BDNF, IL-10 genes in the elderly after 12 weeks of supplementation.
   3. There is an effect of gambier catechin (Uncaria gambir Roxb) supplementation on decreasing plasma MDA levels in the elderly after 12 weeks of supplementation.
3. Research Method Research Design: A randomized controlled trial (RCT) design will be used. Population and Sample:The target population for this study is the elderly aged 60 years and above with mild cognitive impairment (MoCA-INA score of 20-25) residing in Padang City, West Sumatra, Indonesia.
4. Research Procedure

   1. Recruitment and Screening

      1. Participants will be recruited from community centers, senior citizen clubs, and public health facilities in Padang City.
      2. Eligibility criteria will include:

         1. Age 60 years and above
         2. Mild cognitive impairment (MoCA-INA score of 20-25)
         3. No history of neurological or psychiatric disorders
         4. No history of substance abuse or chronic medical conditions that may interfere with cognitive function
         5. Willingness to participate in the study and provide informed consent
   2. Baseline Assessments

   <!-- -->

   1. Demographic information will be collected.
   2. Cognitive function will be assessed using the Montreal Cognitive Assessment-Indonesia (MoCA-INA) test.
   3. Blood samples will be drawn for biochemical analysis, including plasma MDA levels.
   4. Genetic analysis will be conducted to assess the expression of APP, MAPT, BDNF, IL-10, and TGF-β genes.

   c. Intervention
   1. Participants will be randomly assigned to either the intervention or control group.
   2. The intervention group will receive gambier catechin supplementation (Uncaria gambir Roxb) at a daily dose of [Insert dosage] for 12 weeks.
   3. The control group will receive a placebo. d. Follow-up Assessments

   <!-- -->

   1. Cognitive function will be reassessed using the MoCA-INA test at 12 weeks.
   2. Blood samples will be drawn for biochemical analysis and genetic analysis as described in the baseline assessments.
5. Data Analysis

   1. Descriptive statistics will be used to summarize demographic data, cognitive function scores, and biochemical parameters.
   2. Inferential statistics, including t-tests and ANOVA, will be used to compare the differences between the intervention and control groups.
   3. Correlation analysis will be conducted to examine the relationship between cognitive function, genetic expression, and plasma MDA levels.
6. Ethical Considerations

   1. The study will be conducted in accordance with ethical principles and guidelines, including the Declaration of Helsinki.
   2. Informed consent will be obtained from all participants.
   3. Participant confidentiality will be maintained throughout the study.
   4. Any adverse events will be monitored and reported.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 years and above
2. Mild cognitive impairment (MoCA-INA score of 20-25)
3. No history of neurological or psychiatric disorders
4. No history of substance abuse or chronic medical conditions that may interfere with cognitive function
5. Willingness to participate in the study and provide informed consent

Exclusion Criteria:

* Participants who did not take Catechin Capsules for two days in a row

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
To determine the effect of gambir catechin (Uncaria gambir Roxb) supplementation on cognitive function using the MoCA-INA test in the elderly after 12 weeks of supplementation | April to september 2024 ( 6 month)
  scor MoCA: 20 to 25
To determine the effect of gambir catechin (Uncaria gambir Roxb) supplementation on the expression of APP, MAPT, BDNF, IL-10, and TGF-β genes in the elderly after 12 weeks of supplementation. | April to september 2024 ( 6 month)
  Gene expression was measured using PCR
To determine the effect of gambir catechin (Uncaria gambir Roxb) supplementation on plasma MDA levels in the elderly after 12 weeks of supplementation. | April to september 2024 ( 6 month)
  Plasma MDA levels, as a marker of lipid peroxidation, were measured using a UV-vis spectrophotometer and the TBARS assay

CONTACTS AND LOCATIONS:
Overall Officials: Nur Indrawati Lipoeto, Profesor, Principal Investigator — Andalas University
Locations (2):
- Andalas Univercity, Padang, West Sumatera, Fiji
- Andalas Univercity, Padang, West Sumatera, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baba Y, Kaneko T, Takihara T. Matcha consumption maintains attentional function following a mild acute psychological stress without affecting a feeling of fatigue: A randomized placebo-controlled study in young adults. Nutr Res. 2021 Apr;88:44-52. doi: 10.1016/j.nutres.2020.12.024. Epub 2021 Jan 2. PMID 33744591
- [Background] Baba Y, Inagaki S, Nakagawa S, Kaneko T, Kobayashi M, Takihara T. Effects of l-Theanine on Cognitive Function in Middle-Aged and Older Subjects: A Randomized Placebo-Controlled Study. J Med Food. 2021 Apr;24(4):333-341. doi: 10.1089/jmf.2020.4803. Epub 2021 Mar 22. PMID 33751906
- [Background] Ide K, Yamada H, Takuma N, Kawasaki Y, Harada S, Nakase J, Ukawa Y, Sagesaka YM. Effects of green tea consumption on cognitive dysfunction in an elderly population: a randomized placebo-controlled study. Nutr J. 2016 May 4;15(1):49. doi: 10.1186/s12937-016-0168-7. PMID 27142448
- [Background] Baba Y, Inagaki S, Nakagawa S, Kaneko T, Kobayashi M, Takihara T. Effect of Daily Intake of Green Tea Catechins on Cognitive Function in Middle-Aged and Older Subjects: A Randomized, Placebo-Controlled Study. Molecules. 2020 Sep 17;25(18):4265. doi: 10.3390/molecules25184265. PMID 32957612
- See also: Related Info — https://docs.google.com/document/d/1fGb_Y2HUOZUhCwLQSVTtI6m_0FM00qan/edit?usp=sharing&amp;amp;amp;ouid=109214101212266635448&amp;amp;amp;rtpof=true&amp;amp;amp;sd=true
- Available data/document: Analytic Code — https://docs.google.com/spreadsheets/d/1jEVgkxVaewBnQVrAg7jR44Au-PHpsxi-/edit?usp=sharing&amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;ouid=109214101212266635448&amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;rtpof=true&amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;sd=true